CLINICAL TRIAL: NCT02812238
Title: Study to Evaluate the Effect of Nicotinamide Riboside on Immunity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 160129; 16-H-0129
Record Dates: First submitted 2016-06-23; First posted 2016-06-24 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-04-03

CONDITIONS: Atherosclerosis; Diabetes; Coronary Artery Disease
Keywords: Inflammasome; Sirt3; Nicotinamide Riboside; Fasting
MeSH Terms: conditions — Atherosclerosis; Diabetes Mellitus; Coronary Artery Disease; Fasting | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Either NR at 1000mg/day or placebo for one week, followed by a washout period of 2-3 weeks, then a crossover to placebo or NR at 1000mg/day for one additional week. The end point was analyzed at end of each treatment.
  Interventions: Dietary Supplement: Nicotinamide riboside (NR); Drug: Placebo
- Arm 2 (Experimental): Either NR at 1000mg/day or placebo for one week, followed by a washout period of 2-3 weeks, then a crossover to placebo or NR at 1000mg/day for one additional week. The end point was analyzed at end of each treatment.
  Interventions: Dietary Supplement: Nicotinamide riboside (NR); Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide riboside (NR) — NR at dose of 1000mg/day will be given for a period of 7 days in a double blinded fashion either from the start of tx or after 1 week of placebo pills.
Drug: Placebo — Placebo capsule daily for a period of 7 days in a double blinded fashion either from the start of tx or after 1 week of NR at a dose of 1000mg/day.

SUMMARY:
Background:

The immune system controls how the body responds to infection or injury. Researchers want to see what effect a dietary supplement called nicotinamide riboside (NR) has on the immune system. A study showed that fasting has a good effect on immune cell health in healthy people. And when immune cells were exposed to NR they had a similar positive response as with fasting. Researchers want to see if healthy people have the same effects from NR and fasting, and if those effects last.

Objectives:

To see if taking nicotinamide riboside will have the same healthy immune system effects as fasting. To see if these good effects continue even after eating again.

Eligibility:

Healthy volunteers ages 18 - 39 years

Design:

Participants will be screened with medical history, physical exam, and blood tests. Women will have a urine pregnancy test.

Participants will take 4 pills of either NR or a placebo once a day for 1 week.

On day 6, they will not eat or drink anything.

On day 7, they will have a study visit to give a blood sample before and after eating a meal at the clinic.

They will also give a urine sample.

Participants will stop taking the pills for 1 2 weeks.

Participants will take either NR or a placebo once a day for 1 week.

They will repeat day 6 and day 7 of the first week.

Participants will get NR once and placebo once, but will not know which they are taking.

DETAILED DESCRIPTION:
Intermittent caloric restriction or fasting has numerous health effects including the reduction in numerous cardiovascular disease risk factors. The cellular programs activated by caloric restriction are similarly turned on in preclinical studies in response to a 24-hour fast. We have found that a beneficial effect of 24-hour fasting is that it blunts the activation of a component of the immune system, termed the Nod-like receptor family protein 3 (NLRP3) Inflammasome. This inflammasome, as a mediator of sterile inflammation, is associated with the development of diabetes and atherosclerosis. At the same time, we found that refeeding after the 24-hour fast significantly increased NLRP3 protein levels, IL-1Beta, and TNF signaling, and that fasting blunted the NLRP3 inflammasome response, in association with the activation of a fasting sensing protein called SIRT3. Interestingly, a recently discovered naturally occurring form of vitamin B3, called nicotinamide riboside (NR), has been found to activate SIRT3. We found that NR reproduces the NLRP3 inflammasome blunting effect of fasting when administered to primary human monocytes/macrophages in culture. Putting this together, it would be interesting to evaluate whether the administration of NR to human subjects would replicate the fasting blunting effect on the NLRP3 inflammasome. Interestingly, at the same time, it has recently been found, in a preclinical study, that the NLRP3 protein can orchestrate differentiation of naive T- cells into Th2 cells. We therefore propose to more broadly examine the effects of NR administration on myeloid and lymphoid cell biology in healthy volunteers.

ELIGIBILITY:
* INCLUSION CRITERIA:

As this is a pilot study, the age-range and BMI range of subjects will be restricted to potentially reduce metabolic variables associated with a wide age- and BMI-range.

* Males and females between the ages of 18 and 39
* BMI between 18.5 and 29.9
* Agrees to comply with study procedures and maintain current level of physical activity and dietary intake throughout the study.
* Female subjects of child-bearing ability willing to commit to reliable contraception while participating in the study.

EXCLUSION CRITERIA:

* Subjects with an acute or chronic illness as per history, on laboratory analysis or requiring medications to manage disease.
* Subjects taking vitamins or supplements or any medications, except oral contraceptives, within 4 weeks of participation into this study.
* BMI <18.5 or >29.9.
* Female subjects who are pregnant or lactating.
* Subjects who have donated blood or participated in another clinical trial involving blood draws in the last 8 weeks.
* Subjects who use nicotine products including chewing tobacco, vaporizer, gum, cigarette or patch form within three months.
* Any other medical condition that, in the opinion of the Principal Investigator, might put the subject at risk of harm during the study or might adversely affect the interpretation of the study data.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-06-23; Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Sack, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Traba J, Kwarteng-Siaw M, Okoli TC, Li J, Huffstutler RD, Bray A, Waclawiw MA, Han K, Pelletier M, Sauve AA, Siegel RM, Sack MN. Fasting and refeeding differentially regulate NLRP3 inflammasome activation in human subjects. J Clin Invest. 2015 Nov 3;125(12):4592-600. doi: 10.1172/JCI83260. PMID 26529255
- [Background] Canto C, Houtkooper RH, Pirinen E, Youn DY, Oosterveer MH, Cen Y, Fernandez-Marcos PJ, Yamamoto H, Andreux PA, Cettour-Rose P, Gademann K, Rinsch C, Schoonjans K, Sauve AA, Auwerx J. The NAD(+) precursor nicotinamide riboside enhances oxidative metabolism and protects against high-fat diet-induced obesity. Cell Metab. 2012 Jun 6;15(6):838-47. doi: 10.1016/j.cmet.2012.04.022. PMID 22682224
- [Background] Brown KD, Maqsood S, Huang JY, Pan Y, Harkcom W, Li W, Sauve A, Verdin E, Jaffrey SR. Activation of SIRT3 by the NAD(+) precursor nicotinamide riboside protects from noise-induced hearing loss. Cell Metab. 2014 Dec 2;20(6):1059-68. doi: 10.1016/j.cmet.2014.11.003. PMID 25470550
- [Derived] Han K, Singh K, Meadows AM, Sharma R, Hassanzadeh S, Wu J, Goss-Holmes H, Huffstutler RD, Teague HL, Mehta NN, Griffin JL, Tian R, Traba J, Sack MN. Boosting NAD preferentially blunts Th17 inflammation via arginine biosynthesis and redox control in healthy and psoriasis subjects. Cell Rep Med. 2023 Sep 19;4(9):101157. doi: 10.1016/j.xcrm.2023.101157. Epub 2023 Aug 15. PMID 37586364
- [Derived] Wu J, Singh K, Lin A, Meadows AM, Wu K, Shing V, Bley M, Hassanzadeh S, Huffstutler RD, Schmidt MS, Blanco LP, Tian R, Brenner C, Pirooznia M, Kaplan MJ, Sack MN. Boosting NAD+ blunts TLR4-induced type I IFN in control and systemic lupus erythematosus monocytes. J Clin Invest. 2022 Mar 1;132(5):e139828. doi: 10.1172/JCI139828. PMID 35025762
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-H-0129.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotinamide Riboside, Then Placebo: These subjects were first administered Nicotinamide riboside at 1000mg/day or placebo for one week, followed by a washout period of 2-3 weeks, then a crossover to placebo for one additional week.
- Placebo, Then Nicotinamide Riboside: These subjects were first administered Placebo for one week, followed by a washout period of 2-3 weeks, then a crossover to Nicotinamide riboside at 1000mg/day for one week.
Period: First Intervention
Arm/Group | Nicotinamide Riboside, Then Placebo | Placebo, Then Nicotinamide Riboside
Started | 19 | 19
Completed | 18 | 19
Not Completed | 1 | 0
Period: Second Intervention
Arm/Group | Nicotinamide Riboside, Then Placebo | Placebo, Then Nicotinamide Riboside
Started | 18 | 19
Completed | 18 | 18
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: Baseline data for all subjects on the study.
Arm/Group | All Subjects
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 15
  More than one race | 1
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean IL-1 Beta Release From Peripheral Blood Mononuclear Cells During Refeeding After 24 Hour Fast
Description: The IL- 1beta secretion is measured in response to fasting, refeeding and administration of Nicotinamide Riboside (or placebo). Nicotinamide riboside acts as a fasting mimetic, and is supposed to maintain the reduction of IL-1 beta secretion (indicating NLRP3 inflammasome activation) induced by fasting. 1000 mg of Nicotinamide riboside on a daily basis is given to the subjects for a period of 7-10 days.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Nicotinamide Riboside: In this crossover design the study subjects from both arms that had received NR at 1000mg/days/7days, were combined to analyze the effect of NR on IL-1beta secretion in response to refeeding.
- Placebo: In this crossover design the study subjects from both arms that had received placebo for days, were combined to analyze the effect of NR on IL-1beta secretion in response to refeeding.
Arm/Group | Nicotinamide Riboside | Placebo
Number analyzed (Participants) | 36 | 36
mg/dL | 582 (612) | 794 (941)

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Nicotinamide Riboside: These subjects were administered Nicotinamide riboside
- Placebo: These subjects were administered Placebo
Arm/Group | Nicotinamide Riboside | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 3/38 | 2/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nicotinamide Riboside (N=38) | Placebo (N=38)
Headache (General disorders) | 1 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT02812238/Prot_SAP_000.pdf